CLINICAL TRIAL: NCT00636324
Title: Nasal Continuous Positive Airway Pressure in Preterm Infants After Extubation: Comparison of Different Levels of Pressure
Brief Title: Level of Continuous Positive Airway Pressure (CPAP) in Preterm Infants After Extubation (L-CPAP Study)
Acronym: L-CPAP
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Difficulties in recruitment - will require longer time to achieve sample size
Sponsor: Hamilton Health Sciences Corporation (Other)
Responsible Party: Guilherme Mendes Sant'Anna, Hamilton Health Sciences
Organization: McMaster University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REB project # 07-047
Record Dates: First submitted 2008-03-07; First posted 2008-03-14 (Estimated); Last update posted 2009-02-10 (Estimated); Status verified 2009-02

CONDITIONS: Respiratory Insufficiency of Prematurity
Keywords: Respiratory distress syndrome; Preterm infants; Extubation failure; Pneumothorax; Lung injury; Airway pressure
MeSH Terms: conditions — Respiratory Insufficiency; Respiratory Distress Syndrome; Pneumothorax; Lung Injury

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Nasal CPAP, level of 7 to 9 cmH2O
  Interventions: Device: Nasal CPAP, level 7 to 9 cmH2O
- 2 (Active Comparator): Nasal CPAP, level 4 to 6 cmH2O
  Interventions: Device: Nasal CPAP, level 4 to 6 cmH2O

INTERVENTIONS:
Device: Nasal CPAP, level 7 to 9 cmH2O — Apply nasal CPAP pressure of 7-9 H2O for the first 72 hours of extubation
  Other Names: High pressure nCPAP, 7-9 cmH2O
  Arms: 1
Device: Nasal CPAP, level 4 to 6 cmH2O — Apply nasal CPAP pressure of 4 to 6 cmH2O for the first 72 hours of extubation
  Other Names: Low pressure CPAP, 4-6 cmH2O
  Arms: 2

SUMMARY:
Despite widely used of nasal CPAP in preterm infants, uncertainties regarding aspects of its application remain. Clinical indications vary greatly between institutions, especially when combined with varieties of systems, devices, and techniques available. One of the controversial aspects that needs to be clarified is the level of pressure which should be used. The objective of the study is to compare the effectiveness of two ranges of nCPAP pressure that are within the spectrum of current practice for post-extubation support in very preterm infants.

DETAILED DESCRIPTION:
The use of nCPAP has been established as an effective respiratory support to prevent extubation failure and as treatment of other pulmonary diseases. An upsurge in its popularity has resulted in some controversial aspects, including the level of pressure to be used. The level that has been used in very preterm infants after extubation, which mostly came from anecdotal data, varies from 3 to 10 cmH2O.

Physiologic studies show higher nCPAP pressures improve lung mechanical properties. Though potential side effects have been of concern in practical application, there is no formal evidence supporting the concept that increased CPAP pressure results in a higher risk of complications. In relatively stable preterm infants, the range of optimal CPAP level needs to be established in order to adequately support the upper airway and lungs, without increasing complications secondary to the pressure applied. Given the uncertainty of the nCPAP pressure that should be used in very preterm infants, we conduct a randomized controlled trial to compare the effectiveness of two ranges of nCPAP pressure for post-extubation support in very preterm infants.

The purpose of this trial is to compare the rate of successful extubation of using the nasal CPAP level of 7 to 9 cmH2O compared to level of 4 to 6 cmH2O.

ELIGIBILITY:
Inclusion Criteria:

* Birth weight 500 - 1,250 g
* On mechanical ventilation before 7 days of age
* First extubation before 14 days of age

Exclusion Criteria:

* Presence of lethal anomalies or upper airway abnormalities
* IVH, grade 3 or 4
* Neuromuscular disorders
* Receiving muscle relaxation at time of extubation
* Congenital heart disease, except for PDA
* GI problems resulting in a need to avoid gastric distension

Max Age: 14 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 23 (Actual)
Dates: Start 2007-07; Primary Completion 2008-03 (Actual); Study Completion 2010-06 (Estimated)

PRIMARY OUTCOMES:
The rate of successful extubation within 72 hours of extubation | within 72 hours after extubation

SECONDARY OUTCOMES:
The rate of successful extubation within 7 days of extubation | within 14 days after extubation
Number of days on nCPAP | within 14 days after extubation
Occurrence of air leak syndrome | within 14 days after extubation
Occurrence of IVH grade 3 or 4 | within 14 days after extubation
Occurrence of traumatized nasal septum | within 14 days after extubation

CONTACTS AND LOCATIONS:
Overall Officials: Giulherme M SantAnna, MD, Principal Investigator — Hamilton Health Sciences Corporation